CLINICAL TRIAL: NCT03473886
Title: Developing a Positive Psychology Intervention to Promote Health Behaviors in Metabolic Syndrome: Proof-of Concept Trial
Acronym: MAPP-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rachel Millstein, Assistant in Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1K23HL135277-02 (NIH)
Record Dates: First submitted 2018-03-08; First posted 2018-03-22 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm: PP-MI (Experimental): Participants will complete an 8-week group physical activity and positive psychology program, in which they will complete exercises related to increasing positive emotions and physical activity during and between the group sessions. They will track their activity (steps) and set personalized physical activity goals each week, as complete a group walk or indoor exercise during the group sessions. We will ask questions about participants' health and health behaviors, and ask them to wear a physical activity monitor at the beginning and end of the program.
  Interventions: Behavioral: Intervention arm: PP-MI

INTERVENTIONS:
Behavioral: Intervention arm: PP-MI — The positive psychology exercises include gratitude-based activities, strengths-based activities, and meaning-based activities. The physical activity goal setting exercises include the following topics: health benefits, social resources, and neighborhood walkability.

SUMMARY:
Specific Aim #1 (Feasibility; primary aim): To assess the feasibility of the positive psychology (PP)-motivational interviewing (MI) group-based physical activity intervention and outcome assessments in patients with metabolic syndrome (MetS).

Hypothesis: The PP exercises and MI-based goal-setting sessions will be feasible: most (≥50%) of participants will complete 6/8 exercises/sessions. Furthermore, we will be able to obtain objective physical activity measurement follow-up data from at least 80% of enrolled participants at 8 weeks.

Specific Aim #2 (Acceptability): To assess whether the intervention is acceptable to participants, as measured by ratings provided after each PP and MI exercise.

Hypothesis: The intervention will be acceptable: participants will rate each PP and MI exercise with a mean score of at least 7 out of 10 on ratings of ease of completion and helpfulness.

Specific Aim #3 (Outcomes): To assess whether this preliminary intervention appears to result in improvement of physical activity, related health behaviors (sedentary time, diet quality), and psychological well-being (optimism, positive affect, anxiety, depression).

Hypothesis: The intervention will lead to improvements in physical activity, related health behaviors, optimism and positive affect, and reductions in depression and anxiety at 8 weeks compared to baseline.

DETAILED DESCRIPTION:
In this proof-of-concept study, investigators will run two 8-week PP-MI groups (complete n=8 each, n=16 total) for primary care patients with MetS. Investigators will use ratings of feasibility and acceptability for each of the sessions and obtain objective physical activity measures pre- and post- group. Investigators will also obtain questionnaire-based information related to health behavior adherence and psychological and physical health to ensure the feasibility of these methods prior to further testing. Investigators may gather exit interview data to assess participant liking, utility, and additional needs, to allow for further refinement of the intervention.

Baseline information about enrolled participants will be obtained from the patients, care providers, and the electronic medical record as required for characterization of the population. This information will include medical data related to MetS (e.g., blood sugar, blood pressure, body mass index, triglycerides, cholesterol), current medications, and sociodemographic data (age, gender, race/ethnicity, education, marital status).

Participants will attend 90-minute groups sessions that will be held at two primary care clinics (MGH Healthcare Centers). The overall structure of each session will be: 30 minutes for positive psychology exercise review/discussion, 30 minutes for physical activity goal setting, education, and discussion, and 30 minutes for a group walk or indoor exercises in inclement weather.

Participants will be asked to wear an Actigraph GT3x+ accelerometer for 1 week at baseline and 1 week at follow-up to assess the feasibility of doing so. Accelerometers such as this one are considered to be the standard for measuring habitual physical activity. They are pedometer-size devices that attach to a belt and are worn at the waist. Participants will also be given a Fitbit Zip to keep, which they will be asked to wear daily for the duration of the study in order to track their activity (steps).

Upon beginning the groups, participants will be provided with a treatment manual with weekly PP exercises, information about the importance of physical activity and related health behaviors, and how to set goals to improve these behaviors. The PI will lead all groups.

For the first session, in the PP portion, participants will discuss and be assigned the first exercise- gratitude for positive events- and will be instructed to complete the PP exercise during the next week. Prior to completing the exercise, participants will be asked to rate their current levels of happiness and optimism. Immediately after completing the exercise, participants will rate the ease of exercise completion, overall utility of the exercise, and their current levels of happiness and optimism, all using 10-point Likert scales. In the first goal-setting session, we will discuss the importance of physical activity in MetS. Participants will be given a Fitbit Zip to keep, which they will use to track the number of steps they take each day, for the duration of the study. Investigators will review instructions for use and set a goal for monitoring their baseline physical activity over the next week. Fitbits will not be used as an outcome measure but as a tool that participants can use to monitor their activity and set goals. Finally, the last 30 minutes will be spent doing a group walk around the local clinic neighborhood. All group walks and exercises will be done at a pace comfortable for participants.

Participants will be asked to complete the 8 total weekly PP exercises, set physical activity goals, and attend as many group sessions as they can.

All sessions will include (a) a review and discussion of the past week's PP exercise, (b) a discussion of the rationale of the next week's PP exercise using the PP manual, and (c) assignment of the next week's PP exercise. For the goal-setting/MI portion, participants will (a) review their goals and steps from the prior week, (b) discuss techniques for improving physical activity (e.g., monitoring physical activity, taking standing breaks), and (c) set goals for the next week. The exercises and content for both PP and MI will be assigned in the same order for all participants receiving them.

Immediately after the week 8 session, investigators will distribute the same self-report questionnaires that were administered at baseline (before week 1). The Actigraphs will then be collected at this point and the data will be uploaded to assess for valid wear time. If participants have not worn them for enough time (>4 days), investigators will send it home with them and ask them to re-wear it and mail it back.

ELIGIBILITY:
Inclusion Criteria:

• Both of the two MetS components most strongly related to MetS outcomes and most sensitive to lifestyle change:

* elevated abdominal obesity (waist circumference >102 cm in men or >88 cm in women)
* If waist circumference is not available, body mass index (BMI) will be used as a surrogate measure based on prior research (BMI ≥29.1 kg/m2 for men and 27.2 kg/m2 for women).

AND

- elevated blood pressure (systolic ≥130 and/or diastolic ≥85 mm Hg or be on blood pressure medication).

* Plus ≥1 additional MetS component:

  * Serum triglycerides ≥150 mg/dL
  * High-density lipoprotein (HDL) cholesterol <40 mg/dL in men or <50 mg/dL in women
  * Fasting plasma glucose >100mg/dL.
* Suboptimal physical activity defined as ≤150 minutes/week moderate intensity activity, which represents less than national-level recommendations.

Exclusion Criteria:

* Inability to speak/read English
* Cognitive deficits impeding ability to participate or provide informed consent (measured by a 6-item screen)
* Illness likely to lead to death in the next 6 months per PCP
* Current treatment for cancer, liver, or renal disease
* Pregnancy
* Documented severe mental illness (e.g., psychosis, suicidality)
* No telephone access
* Inability to be physically active
* Diabetes or known or suggested cardiac disease, given that this is a primary prevention study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Millstein, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: PP-MI: Participants will complete an 8-week group physical activity and positive psychology program, in which they will complete exercises related to increasing positive emotions and physical activity during and between the group sessions. They will track their activity (steps) and set personalized physical activity goals each week, as they complete a group walk or indoor exercise during the group sessions. We will ask questions about participants' health and health behaviors, and ask them to wear a physical activity monitor at the beginning and end of the program.
  Intervention arm: PP-MI: The positive psychology exercises include gratitude-based activities, strengths-based activities, and meaning-based activities. The physical activity goal setting exercises include the following topics: health benefits, social resources, and neighborhood walk-ability.
Period: Overall Study
Arm/Group | Intervention Arm: PP-MI
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Physical Activity Adherence (Actigraph) [Mean (Standard Deviation); unit: minutes/week] — ActiGraph GT3X+ accelerometers are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer to assess the feasibility of doing so and to ensure adequate capture of physical activity. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  minutes/week
    number analyzed (Participants) | 7
    (all) | 12.5 (10.74)
Life Orientation Test- Revised Scores [Mean (Standard Deviation); unit: score on a scale] — The LOT-R is a well-validated 6-item instrument used to measure dispositional optimism. Higher scores indicate higher levels of optimism. (Range: 5-30) Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 11.7 (2.8)
Positive and Negative Affect Schedule Scores [Mean (Standard Deviation); unit: score on a scale] — The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials, will be used to measure positive affect. Higher scores indicate higher levels of positive affect. (Range: 10-50) Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 36.1 (5.0)
The Hospital Anxiety and Depression Scale - Anxiety Scores Scores [Mean (Standard Deviation); unit: score on a scale] — The HADS will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients. Higher scores indicate higher levels of anxiety. (Range: HADS-A, HADS-D; 0-21 each) Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 6.7 (2.0)
The Neighborhood Environment Walkability Scale-Abbreviated Scores [Mean (Standard Deviation); unit: score on a scale] — NEWS is a 98-question instrument that assesses the perception of neighborhood design features related to physical activity. NEWS-A is an abbreviated version and will be used to measure residents' perceptions of neighborhood design related to physical activity, including places for walking and cycling, aesthetics, traffic hazards, and crime (Range: 16-64). Higher scores indicate greater perceived walkability. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 10.7 (1.6)
Barriers to Being Active Quiz- Lack of Time Scores [Mean (Standard Deviation); unit: score on a scale] — The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the barriers to physical activity. Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of time" category (range of 0-9), and we calculated the score at baseline. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 2.0 (2.5)
The Medical Outcomes Study Short Form-12 Scores - Physical Composite Score [Mean (Standard Deviation); unit: score on a scale] — The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past. (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Baseline scores were calculated. Higher scores indicate higher level of health related QoL. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 41.9 (6.0)
The Community Healthy Activities Model Program for Seniors Scores [Mean (Standard Deviation); unit: minutes per week] — CHAMP is a self-report questionnaire that assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults. It includes activities of various intensities (from light to vigorous) such as walking, running, hiking, swimming, bicycling, dancing, tennis, aerobics, yoga/tai chi, gardening, and housework. The activities are assessed in min/week. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  minutes per week
    number analyzed (Participants) | 7
    (all) | 14.6 (7.7)
Behavioral Risk Factor Surveillance System Fruit and Vegetable Module - Fruit Category [Mean (Standard Deviation); unit: fruits/day] — The CDC's BRFSS Fruit and Vegetable Module is a brief questionnaire about frequency of eating different types of fruits and vegetables. It assesses the frequency of consumption of 100% fruit juice, fruit, beans (legumes), dark green vegetables, orange vegetables, and other vegetables over the past month. The outcome measure is the number of fruits consumed per day. Population: Although 8 participants were enrolled in the study, 6 participants completed this specific measure at the baseline assessment.
  fruits/day
    number analyzed (Participants) | 6
    (all) | 1.2 (1.5)
National Cancer Institute's Percentage Energy from Fat Screener Scores [Mean (Standard Deviation); unit: number of times consumed per day] — The National Cancer Institute's Percentage Energy from Fat Screen is a brief questionnaire that estimates people's typical percentage of energy derived from eating common fat-containing foods, as fat content is related to metabolic syndrome progression. The questionnaire converts an individual's responses to an estimate of that individual's percentage energy from fat. Higher scores indicate higher fat consumption. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  number of times consumed per day
    number analyzed (Participants) | 7
    (all) | 3.9 (2.8)
HADS-D Scores [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients.(Range: 0-21). Baseline scores were calculated. Higher scores indicate worse outcome (i.e. greater levels of depression). Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 4.6 (2.9)
Barriers to Being Active Quiz Score- Social Influence [Mean (Standard Deviation); unit: score on a scale] — The BBAQ is a 21-item measure that assesses barriers to physical activity. The domain, social influence, contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores the "social influence" category (range of 0-9), and we calculated the baseline score. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 3.4 (2.3)
Barriers to Being Active Quiz Score- Lack of Energy [Mean (Standard Deviation); unit: score on a scale] — The BBAQ is a 21-item measure, assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of energy" category (range of 0-9), and we calculated the score at baseline. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 1.3 (2.6)
Barriers to Being Active Quiz Score- Lack of Willpower [Mean (Standard Deviation); unit: score on a scale] — The BBAQ is a 21-item measure, assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of will power" category (range of 0-9), and we calculated the score at baseline. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 5.9 (0.7)
Barriers to Being Active Quiz Score - Fear of Injury [Mean (Standard Deviation); unit: score on a scale] — The BBAQ is a 21-item measure assesses the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "fear of injury" category (range of 0-9), and we calculated the score at baseline. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 1.4 (1.6)
Barriers to Being Active Quiz Score - Lack of Skill [Mean (Standard Deviation); unit: score on a scale] — The BBAQ is a 21-item measure that assesses the barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of skill" category (range of 0-9), and we calculated the score at baseline. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 2.7 (0.6)
Barriers to Being Active Quiz Score - Lack of Resources [Mean (Standard Deviation); unit: score on a scale] — The BBAQ is a 21-item measure that assesses the barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of resources" category (range of 0-9), and we calculated the score at baseline. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 2.7 (2.8)
SF-12 Scores - Mental Composite Score [Mean (Standard Deviation); unit: score on a scale] — The Medical Outcomes Study Short Form-12 (SF-12) was used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past. (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Higher scores indicate higher level of health related QoL. Population: Although 8 participants were enrolled in the study, 7 participants completed this specific measure at the baseline assessment.
  score on a scale
    number analyzed (Participants) | 7
    (all) | 48.2 (8.2)
BRFSS- Vegetable Module [Mean (Standard Deviation); unit: vegetable/day] — The CDC's BRFSS Fruit and Vegetable Module is a brief questionnaire about frequency of eating different types of fruits and vegetables. It assesses the frequency of consumption of 100% fruit juice, fruit, beans (legumes), dark green vegetables, orange vegetables, and other vegetables over the past month. The outcome measure is the number of vegetables consumed per day. Population: Although 8 participants were enrolled in the study, 6 participants completed this specific measure at the baseline assessment.
  vegetable/day
    number analyzed (Participants) | 6
    (all) | 1.5 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of PP-MI-Based Health Behavior Intervention Exercises Completed
Description: Feasibility will be measured by examining the number of completed exercises.
Time Frame: 8 weeks of group sessions
Measure: Mean (Standard Deviation); unit: Exercises completed
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
Exercises completed | 7.0 (0.5)

2. Primary Outcome: Number of Participants Completing Objective Physical Activity Measurement
Description: Feasibility will be measured by examining the number of participants who wore Actigraphs with sufficient wear time both at baseline and at follow-up
Time Frame: 8 weeks of group sessions
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
Participants | 7

3. Secondary Outcome: Acceptability of Intervention
Description: Acceptability of the intervention was assessed through participants' ratings of each PP and MI exercise. Participants will provide ratings of utility after each exercise, measured on a 10-point Likert scale (0=not at all helpful;10=very helpful). Weekly utility ratings were averaged to provide an overall utility score of the exercises.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale | 8.1 (1.0)

4. Secondary Outcome: Physical Activity Adherence (Actigraph)
Description: ActiGraph GT3X+ accelerometers are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer to assess the feasibility of doing so and to ensure adequate capture of physical activity.
Time Frame: Change in physical activity level from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
minutes/week
  Baseline | 12.5 (10.74)
  Week 8 | 40.9 (70.6)

5. Secondary Outcome: Changes in Life Orientation Test- Revised Scores
Description: Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism. (Range: 0-24) Change was calculated by subtracting the score at baseline from the score at 8 weeks. Higher scores indicate higher levels of optimism.
Time Frame: Change in dispositional optimism from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 11.7 (2.8)
  8 Weeks | 10.1 (3.1)

6. Secondary Outcome: Changes in Positive and Negative Affect Schedule Scores
Description: The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect. (Range: 10-50). Change was calculated by subtracting the score at baseline from the score at 8 weeks. Higher scores indicate higher levels of positive affect.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 36.1 (5.0)
  8 Weeks | 40.7 (5.3)

7. Secondary Outcome: Changes in The HADS-A Scores
Description: The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients. (Range:0-21) Change was calculated by subtracting the score at baseline from the score at 8 weeks. Higher scores indicate higher levels of anxiety.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 6.7 (2.0)
  8 Weeks | 5.6 (2.8)

8. Secondary Outcome: Changes in The Neighborhood Environment Walkability Scale-Abbreviated Scores
Description: Measure Description: NEWS is a 98-question instrument that assesses the perception of neighborhood design features related to physical activity. NEWS-A is an abbreviated version and will be used to measure residents' perceptions of neighborhood design related to physical activity, including places for walking and cycling, aesthetics, traffic hazards, and crime (Range: 16-64). Higher scores indicate greater perceived walkability.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 10.7 (1.6)
  8 Weeks | 10.8 (1.8)

9. Secondary Outcome: Changes in Barriers to Being Active Quiz- Lack of Time Scores
Description: The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of time" category (range of 0-9), and we calculated the change in score from baseline to 8 weeks.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 2.0 (2.5)
  8 Weeks | 2.3 (2.0)

10. Secondary Outcome: Changes in The Medical Outcomes Study Short Form-12 Scores - Physical Composite Score
Description: The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past. (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Change was calculated by subtracting the score at baseline from the score at 8 weeks. Higher scores indicate higher level of health related QoL.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 41.9 (6.0)
  8 Weeks | 44.6 (9.9)

11. Secondary Outcome: Changes in The Community Healthy Activities Model Program for Seniors Scores
Description: CHAMP is a self-report questionnaire that assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults. It includes activities of various intensities (from light to vigorous) such as walking, running, hiking, swimming, bicycling, dancing, tennis, aerobics, yoga/tai chi, gardening, and housework. The activities are assessed in min/week.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
minutes per week
  Baseline | 14.6 (7.7)
  8 Weeks | 23.1 (3.6)

12. Secondary Outcome: Changes in Behavioral Risk Factor Surveillance System Fruit and Vegetable Module - Fruit Category
Description: Measure Description: The CDC's BRFSS Fruit and Vegetable Module is a brief questionnaire about frequency of eating different types of fruits and vegetables. It assesses the frequency of consumption of 100% fruit juice, fruit, beans (legumes), dark green vegetables, orange vegetables, and other vegetables over the past month. The outcome measure is the number of fruits consumed per day.
Time Frame: Change in # of fruits consumed/day from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: fruits/day
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 6
fruits/day
  Baseline | 1.2 (1.5)
  8 Weeks | 1.1 (0.9)

13. Secondary Outcome: Changes in National Cancer Institute's Percentage Energy From Fat Screener Scores
Description: The National Cancer Institute's Percentage Energy from Fat Screen is a brief questionnaire that estimates people's typical percentage of energy derived from eating common fat-containing foods, as fat content is related to metabolic syndrome progression. The questionnaire converts an individual's responses to an estimate of that individual's percentage energy from fat. Higher scores indicate higher fat consumption.
Time Frame: Change in number of times fat is consumed per day from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: # of times fat consumed/day
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
# of times fat consumed/day
  Baseline | 3.9 (2.8)
  8 Weeks | 3.4 (1.1)

14. Secondary Outcome: Change in HADS-D Scores
Description: The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients.(Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 8 weeks. Higher scores indicate worse outcome (i.e. greater levels of depression).
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 4.6 (2.9)
  8 Weeks | 2.4 (1.8)

15. Secondary Outcome: Change in Barriers to Being Active Quiz Score- Social Influence
Description: The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "social influence" category (range of 0-9), and we calculated the change in score from baseline to 8 weeks.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 3.4 (2.3)
  8 Weeks | 2.3 (1.9)

16. Secondary Outcome: Change in Barriers to Being Active Quiz Score- Lack of Energy
Description: The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of energy" category (range of 0-9), and we calculated the change in score from baseline to 8 weeks.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 1.3 (2.6)
  8 Weeks | 1.9 (2.0)

17. Secondary Outcome: Change in Barriers to Being Active Quiz Score- Lack of Willpower
Description: The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of will power" category (range of 0-9), and we calculated the change in score from baseline to 8 weeks.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 5.9 (0.7)
  8 Weeks | 2.1 (1.3)

18. Secondary Outcome: Change in Barriers to Being Active Quiz Score - Fear of Injury
Description: The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "fear of injury" category (range of 0-9), and we calculated the change in score from baseline to 8 weeks.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 1.4 (1.6)
  8 Weeks | 1.1 (1.2)

19. Secondary Outcome: Change in Barriers to Being Active Quiz Score - Lack of Skill
Description: The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of skill" category (range of 0-9), and we calculated the change in score from baseline to 8 weeks.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 2.7 (0.6)
  8 Weeks | 1.1 (1.2)

20. Secondary Outcome: Change in Barriers to Being Active Quiz Score - Lack of Resources
Description: The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely." This outcome explores "lack of resources" category (range of 0-9), and we calculated the change in score from baseline to 8 weeks.
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 2.7 (2.8)
  8 Weeks | 1.4 (1.3)

21. Secondary Outcome: Change in SF-12 Scores - Mental Composite Score
Description: as for outcome 10
Time Frame: Change in score from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 7
score on a scale
  Baseline | 48.2 (8.2)
  8 Weeks | 54.2 (8.2)

22. Secondary Outcome: Change in BRFSS- Vegetable Module
Description: Measure Description: The CDC's BRFSS Fruit and Vegetable Module is a brief questionnaire about frequency of eating different types of fruits and vegetables. It assesses the frequency of consumption of 100% fruit juice, fruit, beans (legumes), dark green vegetables, orange vegetables, and other vegetables over the past month. The outcome measure is the number of vegetables consumed per day.
Time Frame: Change in # of vegetables consumed/day from Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: vegetable/day
Arm/Group | Intervention Arm: PP-MI
Number analyzed (Participants) | 6
vegetable/day
  Baseline | 1.5 (0.8)
  8 Weeks | 1.9 (0.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events are "any untoward or unfavorable medical occurrence in a human subject including any abnormal sign, symptom or disease...whether or not associated with the subject's participation in the research."
Arm/Group | Intervention Arm: PP-MI
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm: PP-MI (N=8)
Pain after walking (Musculoskeletal and connective tissue disorders) | 1 (1) — The participant reported an exacerbation of her existing condition (baker's cyst) on a day when she overpaced herself with walking. She rested the next day, used a knee brace until the pain relieved, and did not require other additional assistance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03473886/Prot_SAP_000.pdf